CLINICAL TRIAL: NCT00775892
Title: A Multi-Center Open Label Study to Evaluate the SeriACL™ Device (Gen IB) for Primary Anterior Cruciate Ligament Repair
Brief Title: SeriACL™ Device (Gen IB) Trial for Anterior Cruciate Ligament (ACL) Repair
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Serica Technologies, Inc. (Industry)
Responsible Party: Rebecca L Horan, PhD, Serica Technologies, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-ACL1B
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: ACL; Ligament

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: SeriACL Device ACL Reconstruction — Long-term Bioresorbable ACL Scaffold

SUMMARY:
A multi-center single-arm clinical trial is being conducted to evaluate SeriACL device safety and performance during total anterior cruciate ligament (ACL) reconstruction.

ELIGIBILITY:
Major Inclusion Criteria:

* Complete rupture of the ACL
* Passive flexion >= 120° and passive extension = contralateral knee
* MCL grade 2 or less
* Pre-injury Tegner score >= 4
* Informed Consent

Major Exclusion Criteria:

* Prior ACL reconstruction.
* Severe pain, swelling, or redness
* Complete PCL tear
* Complex menisci tears
* Contralateral knee ligament injury
* OA > Grade II

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety - Adverse Events | 12 months
KT-1000 Arthrometer Knee Laxity | 12 months

SECONDARY OUTCOMES:
Knee Surveys | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans Paessler, MD, Principal Investigator — ATOS Clinic, Heidelberg; Johan Bellemans, MD, Principal Investigator — UZ Leuven, Belgium; Holger Schmitt, MD, Principal Investigator — Heidelberg University; Gerhard Oberthaler, MD, Principal Investigator — Dr. Pierer Sanatorium, Salzburg, Austria; Uwe Pietzner, MD, Principal Investigator — Dietrich-Bonhöffer-Klinik, Altentreptow, Germany; Michael Jagodzsinki, MD, Principal Investigator — Hannover Medical School
Locations (6):
- Dr. Pierer Sanatorium, Salzburg, Austria
- UZ Leuven, Leuven, Belgium
- Germany (4):
  - Dietrich-Bonhöffer-Klinik, Altentreptow
  - Medizinische Hochschule Hannover, Hanover
  - ATOS Clinic, Heidelberg
  - University of Heidelberg, Heidelberg